CLINICAL TRIAL: NCT03411577
Title: Development and Testing of a Jamaican Mother-daughter HIV Risk-reduction Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston College (Other)
Collaborators: University of the West Indies, Mona Campus, Kingston, Jamaica (Unknown); University of Pennsylvania (Other); New York University (Other)
Responsible Party: Principal Investigator, Mary Katherine Hutchinson, Professor, Boston College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R01NR010478 (NIH)
Record Dates: First submitted 2018-01-03; First posted 2018-01-26 (Actual); Last update posted 2018-01-26 (Actual); Status verified 2018-01

CONDITIONS: Parent-Child Relations; HIV Prevention; Adolescent Behavior
MeSH Terms: conditions — Adolescent Behavior | interventions — Behavior Therapy

STUDY DESIGN:
Intervention Model Description: Mother-daughter dyads were randomly assigned to either HIV risk-reduction intervention group or control group
Who Masked: Outcomes Assessor
Masking Description: Data collectors were unaware of group assignment of participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavioral Intervention (Experimental): The adolescent HIV/STI risk-reduction intervention aims to: (a) increase knowledge of HIV risk and prevention; (b) strengthen behavioral beliefs regarding abstinence and safer sex; (c) increase self-efficacy and intentions to avoid unsafe sex; and (d) increase sexual communication and refusal skills. The mother component includes much of the same prevention knowledge and addresses parent-teen sexual risk communication, monitoring, and sexual role modeling. Interventions are held on two consecutive Saturdays for 6 hours each day. Mothers' groups meet separately from daughters' groups, although the groups will come together for the last module of each day.
  Interventions: Other: Behavioral Intervention
- Control Group (No Intervention): The control / comparison group is essentially a "no intervention / wait-list" control group. However, during pilot testing, participants expressed a strong desire to engage in some type of health activity. As a result, the control group members, both mothers and daughters, participated in a brief educational activity on reducing risk for cardiovascular disease. The educational activity was limited to a few hours on one Saturday. Participants returned the following week to complete post-test questionnaires along with the participants in the experimental group.

INTERVENTIONS:
Other: Behavioral Intervention
  Arms: Behavioral Intervention

SUMMARY:
Caribbean nations, including Jamaica, exhibit HIV rates that are second only to sub-Saharan Africa. Jamaican young women and adolescent girls are at particularly high risk due to a number of cultural factors, gender norms, partnering with older male partners, and lack of knowledge and skills related to sexual refusal and HIV prevention. U.S. studies have shown that mothers may act as a key influence of their daughters' sexual risk beliefs and behaviors. However, no such studies have documented these effects outside of the U.S. and no studies have evaluated HIV risk-reduction interventions with Jamaican adolescent girls and their mothers. Hence, the purpose of this study is to partner with the University of the West Indies, Jamaican community based organizations (CBOs) and families in order to develop and test a culture-specific mother-daughter HIV risk-reduction intervention in a randomized field experiment. Specifically, the investigative team will evaluate whether a culture-specific, theory-based, skill-building intervention with Jamaican adolescent girls and their mothers can directly and/or indirectly reduce these girls' HIV risk-associated sexual behaviors. Jamaican girls, ages 13 - 17, and their mothers/female guardians will be recruited from CBOs and randomly assigned to either: (a) a mother-daughter HIV risk-reduction intervention condition or (b) a "no intervention" waitlist control condition. The HIV risk-reduction intervention includes 12 1-hour modules scheduled over 2 days and implemented by trained adult Jamaican women (nurses and CBO staff). The mother component is designed to increase those parenting behaviors (e.g., monitoring and parent-teen sexual risk communication [PTSRC]) associated with reduced adolescent sexual risk-taking; the teen component is designed to improve girls' beliefs and skills related to abstinence, sexual negotiation and condom use. A "waitlist" control condition is being employed as the proposed project is a pilot study of the HIV risk-reduction intervention. Primary outcomes include mothers'/daughters' reports of parenting behaviors (monitoring and PTSRC) and daughters' self-reports of sexual risk behaviors (sexual intercourse, unprotected sex, condom use, number of partners). Secondary outcomes include daughters' STI rates, mothers' beliefs regarding parenting behaviors and daughters beliefs regarding sexual risk behaviors.

DETAILED DESCRIPTION:
Caribbean nations, including Jamaica, exhibit HIV rates that are second only to sub-Saharan Africa. Jamaican young women and adolescent girls are at particularly high risk for HIV and other sexually transmitted infections (STIs) due to a number of cultural factors (including male-dominated gender norms and older male partners) and lack of knowledge and skills related to sexual communication, refusal and HIV prevention. Reducing the sexual risk behaviors of Jamaican adolescent females is critical to reducing their risk for HIV/STIs. U.S. studies have shown that parents, particularly mothers, may act as key influences of their daughters' sexual risk beliefs and behaviors. However, no studies have documented these parental effects outside of the U.S. and no studies have evaluated the effectiveness of family-based HIV risk-reduction interventions with international populations, including Jamaican adolescents. Further, it is not yet known whether the instruments used to assess the theoretical constructs of interest are culturally sensitive or appropriate for use with Jamaican adolescents and adults. Hence, the broad objective of this proposal is to develop and test a culturally sensitive, theory-based, gender-specific Jamaican mother-daughter HIV risk-reduction intervention by using community-based participatory research methods and existing collaborative relationships between investigators from the New York University, the University of Pennsylvania Center for Health Disparities Research (PENN) and the University of the West Indies (UWI), Mona Campus. Building upon already completed preliminary elicitation research with Jamaican adolescents, parents, teachers and stakeholders, the investigative team proposes to a) conduct in-depth elicitation research into the social, cultural and family factors that influence HIV-related sexual risk behaviors among Jamaican adolescent girls; b) collaboratively develop a culturally appropriate, gender specific, theory-based mother-daughter HIV risk reduction intervention for Jamaican adolescent girls and their mothers; c) enhance the research capacity of the UWI School of Nursing and the sustainability of the intervention program; d) assess the cultural appropriateness of study instruments and adapt and refine as needed; and e) evaluate the effectiveness of the mother-daughter HIV/STI risk reduction intervention through a randomized pilot study. Although the term "mother" is used throughout the application, it is defined based upon the preliminary elicitation research already completed in Jamaica. The term "mother" will be used to represent the primary female guardian or caregiver; this may be the mother, step-mother, aunt, grandmother or other related or unrelated female guardian or caregiver. In the proposed pilot study, the plan is to recruit 360 Jamaican adolescent females, ages 13 - 17 years, and their mothers from non-governmental community-based organizations (CBOs) in and around Kingston, Jamaica and randomly assign them to either a mother-daughter HIV/STI risk-reduction intervention condition or a "no intervention" waitlist control condition that includes only a brief educational activity addressing heart disease. The HIV risk-reduction intervention will be implemented by trained adult Jamaican women (nurses and CBO staff). The adolescent component is designed to reduce HIV-related sexual risk behaviors (e.g., sexual intercourse, unprotected intercourse, multiple partners); the mother component is designed to increase those parenting behaviors (e.g., monitoring and parent-teen sexual risk communication [PTSRC]) associated with reduced adolescent sexual risk-taking. A "no intervention" waitlist control condition is being employed as the proposed project is a pilot study of the HIV/STI risk-reduction intervention. Should the pilot study find evidence of intervention effectiveness, a full RCT study with long-term follow-up and examination of moderation of intervention effects will be proposed in a subsequent application.

There are four specific aims for the proposed project. Aim 1 is to conduct broad, in-depth elicitation research using community-based participatory research (CBPR) methods in order to elucidate the social, cultural and family factors that influence Jamaican adolescent girls' sexual risk-taking during Years 01 and 02. Aim 2 is to develop a culturally appropriate, gender specific, theory-based, skill-building mother-daughter HIV/STI risk-reduction intervention during Year 02. Aim 3 is to evaluate the cultural appropriateness of our commonly used measures and research instruments using both qualitative and quantitative methods in Year 02. The remaining Aims evaluate the effectiveness of the Jamaican Mother-Daughter HIV/STI Risk-Reduction Project through a randomized pilot study. Aim 4A is to examine whether mothers in the HIV/STI risk-reduction intervention condition show a greater increase in intentions and actual parenting behaviors (monitoring and PCSC) at 3- and 6-month follow-ups compared with mothers in the control group. Aim 4B is to examine whether adolescent girls in the HIV/STI risk-reduction intervention condition show a greater increase in intentions and reduction in actual sexual risk behaviors (sexual intercourse, unprotected intercourse, number of sexual partners) at 3- and 6-month follow-ups compared with girls in the control group. Aim 4C is to examine whether adolescents in the HIV/STI risk-reduction intervention exhibit a lower incidence of clinically documented STIs at 6-month follow-up compared with the adolescents in the control condition. Aim 4D is to identify why and how the mother-daughter HIV/STI risk-reduction intervention works (i.e., mediation of effects). The mother-daughter intervention is based on a family expansion of the Theory of Planned Behavior. The intervention is intended to affect the adolescents' sexual risk behaviors (abstinence, intercourse, unprotected intercourse, condom use, number of partners) by affecting their behavioral, normative and control beliefs and intentions toward safer sex and sexual risk behaviors. It is also designed to affect mothers' key parenting behaviors (monitoring and PTSRC) by affecting their behavioral beliefs, normative beliefs, control beliefs, and intentions toward those parenting behaviors. Parenting behaviors should, in turn, indirectly affect adolescents' sexual risk beliefs, intentions and behaviors. Thus, these theoretical mediators will be assessed in order to understand why the intervention is effective or not. Findings from this study will contribute to the development of effective HIV/STI risk-reduction programs for Jamaican adolescent girls. Significant information will also be gained regarding the design of effective family-based interventions, how to partner with international organizations and communities, and how to develop culturally appropriate instruments and effective HIV risk-reduction interventions for use with international populations at highest risk for HIV/AIDS.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for the adolescent include:

* age between 13- to 17-years, inclusive
* resident of one of the three parishes in and around Kingston, Jamaica (the study area)
* plan to reside in the "study area" for the next 12 months
* able to read, write and understand English
* unmarried and
* agrees to participate and
* mother or primary female guardian also agrees to participate.

Inclusion criteria for the mother/female guardian include:

* age greater than 18
* resident of one of the three parishes in and around Kingston, Jamaica (the study area)
* plan to reside in the "study area" for the next 12 months
* able to read, write and understand English and
* agrees to participate

Exclusion Criteria:

* adolescent and/or mother who is/are disruptive and/or otherwise unable to participate in small group intervention activities
* adolescent who is married

Ages: 13 Years to 17 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 662 (Actual)
Dates: Start 2007-09-29 (Actual); Primary Completion 2011-07-28 (Actual); Study Completion 2012-06-30 (Actual)

PRIMARY OUTCOMES:
Change in adolescent girls' baseline self-reported frequency of condom use at 3 and 6 months | Assessed at baseline, 3- and 6-months; reported for past 3 months
  Questionnaire - self-reported single item asking frequency of condom use during past 3 months; scores range from 1 - 5; higher scores indicate greater frequency of condom use

SECONDARY OUTCOMES:
Adolescent girls' clinically documented STIs | Assessed at baseline and 6-month follow-up
  Urine pcr tests for chlamydia and gonorrhea
Change in adolescent girls' baseline self-reported condom use intentions at 3 and 6 months | Assessed at baseline, 3- and 6-months; reported for next 3 months
  Questionnaire - self-reported single item asking intentions to use condoms during next 3 months; scores range from 1 to 5; higher scores indicate greater intentions
Change in adolescent girls' baseline HIV knowledge scale scores at 3 and 6 months | Assessed at baseline and 3- and 6-month follow-up
  Questionnaire - HIV/AIDS Knowledge Scale - 19 items; scores range from 0 - 19 with higher scores indicating greater amounts of knowledge
Changes in mothers' baseline HIV knowledge scale scores at 3 and 6 months | Assessed at baseline and 3- and 6-month follow-up
  Questionnaire - HIV/AIDS Knowledge Scale - 19 items; scores range from 0 - 19 with higher scores indicating greater amounts of knowledge
Change in mothers' baseline parental monitoring scale scores at 3 and 6 months | Assessed at baseline and 3- and 6-month follow-up; reported for past 3 months
  Questionnaire - self-reported 10-item scale of parental monitoring reported by daughters ; total scores range from 10 - 50; higher scores indicate more parental monitoring/supervision
Change in adolescent girls' baseline parent-teen sexual risk communication (PTSRC) scale scores at 3 and 6 months | Assessed at baseline and 3- and 6-month follow-up; reported for past 3 months
  Questionnaire - PTSRC-III scale; 8 items; total scores range from 5 - 40; higher scores indicate greater sexual communication

CONTACTS AND LOCATIONS:
Overall Officials: Mary K Hutchinson, PhD, Principal Investigator — Boston College

IPD SHARING:
Plan to Share IPD: Undecided
Decisions regarding data sharing will be made on a case-by-case basis. Those who would like to request data should contact the principal investigator.

REFERENCES:
- [Background] Hutchinson MK, Smith TK, Waldron N, Kahwa E, Hewitt HH, Hamilton PI, Kang SY. Validation of the Jamaican Maternal Sexual Role Modelling Questionnaire. West Indian Med J. 2012 Dec;61(9):897-902. doi: 10.7727/wimj.2011.198. PMID 24020230
- [Background] Waldron, N., Hutchinson, M.K., Hewitt, H., Kahwa, E., & Hamilton, P. (2012). Cross-cultural psychometric assessment of the parent-teen sexual risk communication scale in Jamaica. Open Journal of Preventive Medicine, 2(2), 205-213
- [Background] Hutchinson MK, Wood EB. Reconceptualizing adolescent sexual risk in a parent-based expansion of the Theory of Planned Behavior. J Nurs Scholarsh. 2007;39(2):141-6. doi: 10.1111/j.1547-5069.2007.00159.x. PMID 17535314
- [Background] Ajzen, I. (1991). The theory of planned behavior. Organizational Behavior and Human Decision Processes, 50, 179-211.
- [Background] Hutchinson MK. The Parent-Teen Sexual Risk Communication Scale (PTSRC-III): instrument development and psychometrics. Nurs Res. 2007 Jan-Feb;56(1):1-8. doi: 10.1097/00006199-200701000-00001. PMID 17179868
- [Result] Hutchinson MK, Jemmott LS, Wood EB, Hewitt H, Kahwa E, Waldron N, Bonaparte B. Culture-specific factors contributing to HIV risk among Jamaican adolescents. J Assoc Nurses AIDS Care. 2007 Mar-Apr;18(2):35-47. doi: 10.1016/j.jana.2007.01.008. PMID 17403495
- [Result] Kang SY, Hutchinson MK, Waldron N. Characteristics related to sexual experience and condom use among Jamaican female adolescents. J Health Care Poor Underserved. 2013 Feb;24(1):220-32. doi: 10.1353/hpu.2013.0023. PMID 23377730
- [Result] Hutchinson MK, Kahwa E, Waldron N, Hepburn Brown C, Hamilton PI, Hewitt HH, Aiken J, Cederbaum J, Alter E, Sweet Jemmott L. Jamaican mothers' influences of adolescent girls' sexual beliefs and behaviors. J Nurs Scholarsh. 2012 Mar;44(1):27-35. doi: 10.1111/j.1547-5069.2011.01431.x. Epub 2012 Feb 16. PMID 22339731